CLINICAL TRIAL: NCT05188755
Title: Fitness Assessment in Young Adults Recovered From Lymphoma or Hodgkin's Disease
Brief Title: Fitness Assessment in Young Adults Recovered From Lymphoma
Acronym: CUPCAKE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: RBHP 2021 KANOLD; 2021-A02184-37 (Other: ANSM)
Record Dates: First submitted 2021-11-29; First posted 2022-01-12 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2021-11

CONDITIONS: Young Adults; Lymphoma, Non-Hodgkin; Hodgkin Disease
Keywords: physical fitness; fat oxidation; metabolism; exercise
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Hodgkin Disease; Motor Activity | interventions — Cardiac Output; Body Composition; Hematologic Tests; Accelerometry

STUDY DESIGN:
Intervention Model Description: group 1: healthy controls group 2 : young adults recovered from lymphoma or Hodgkin's disease
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy controls (Active Comparator): sex and age matched healthy controls
  Interventions: Other: Indirect calorimetric test during submaximal exercise
- young adults recovered from lymphoma or Hodgkin's disease (Experimental): young adults recovered from lymphoma or Hodgkin's disease
  Interventions: Other: Indirect calorimetric test during submaximal exercise

INTERVENTIONS:
Other: Indirect calorimetric test during submaximal exercise — * metabolic evaluation by indirect calorimetry at rest and during exercise
  * evaluation of cardiac output
  * peripheral quantitative computed tomography (pQCT) of the muscle cross section
  * evaluation of body composition
  * assessment of physical capacity (chair test and 3 min step-test)
  * blood test
  * assess the level of physical activity
  Other Names: cardiac output; body composition; assessment of physical capacity; blood test; accelerometry; peripheral quantitative computed tomography

SUMMARY:
Regular physical activity (PA) is associated with maintaining body composition, increased cardiorespiratory capacity, muscle mass and bone mineral density. In the event of a cancer, the development of physical capacities and metabolism may therefore be disturbed by cancer, these associated treatments (chemotherapy, radiotherapy and hematopoietic stem cell transplantation) but also undernutrition and the reduction in physical activity or even a sedentary lifestyle.

Although the benefits of PA in oncology are now well identified for adult populations, studies are still rare in the population of children, adolescents and young adults, and the results are still difficult to generalize. As a result, there is no recommendation on the practice of physical activity in pediatric oncology or adolescents and young adults and the levels of physical activity of cured patients remain lower than those of the general population.

Fitness is a marker of health in adults as well as in adolescents. Physical condition is a set of components such as cardiorespiratory capacity (transport and use of O2), body composition (distribution of bone, muscle and fat masses) and muscle function (strength, power, fatigue, energy metabolism) .

The investigators hypothesize that, compared to young adults, recovered from lymphoma are expected to exhibit impaired physical condition, due to physical deconditioning.

ELIGIBILITY:
Inclusion Criteria:

* Young adult male or female, aged 18 to 25
* giving free and informed consent
* Hodgkin lymphoma or non-Hodgkin lymphoma in the healing stage
* Cured (defined by an undetectable disease at the end of treatment) for at least one year and maximum 6 years of lymphoma or Hodgkin's disease

Exclusion Criteria:

* Legal incapable adults
* People under judicial protection
* Treatment with systemic glucocorticoids for more than a week, during the 30 days preceding the tests
* Medical contraindication to the practice of physical exercise
* Any pathologies (other than the history of lymphoma for the cases) likely to affect the metabolism or the muscle mass
* Any treatment that may have an influence on the energy metabolism
* Active infection
* Pregnant, breastfeeding, or likely to be
* Subject's refusal to participate

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-06 (Actual); Study Completion 2022-12-06 (Actual)

PRIMARY OUTCOMES:
fat oxidation rate | day at 11:30 am during one day
  maximum rate of lipid oxidation (in mg/ml)

SECONDARY OUTCOMES:
rest metabolism | at 08:00 am in fasted condition during one day
  energy expenditure at rest in kcal.
blood insulinemia | at 07:30 am in fasted condition during one day
  blood value of insulin in pmol/L
blood N-terminal pro-B natriuretic peptide | at 07:30 am in fasted condition during one day
  blood N-terminal pro-B natriuretic peptide level in g/L
blood troponin | at 07:30 am in fasted condition during one day
  blood troponin level in g/L
blood lipids | at 07:30 am in fasted condition during one day
  blood lipids level in g/L
blood glucose | at 07:30 am in fasted condition during one day
  blood glucose level in g/L
Body composition: fat | at 07:30 am during one day
  percentage of fat
Body composition: lean mass | at 07:30 am during one day
  percentage of lean mass
cardiac output | at 11:30 am during one day
  Systolic Ejection Volume in mL evaluated at rest and during submaximal exercise
peripheral quantitative computed tomography | at 10:45 am during one day
  Cross-sectional area of thigh muscles and intermuscular adipose tissue were assessed for muscle at 40% of the length between the greater trochanter and the mid-patella of the right leg
physical condition | at 08:45 am during one day
  3 min step-test (number of ascent / descent step)
physical capacity | at 08:45 am during one day
  chair test (time in second held in position)
physical activity level | from day 2 to day 5
  daily energy expenditure (in Kcal)
sedentary level | from day 2 to day 5
  total sedentary time (in min) evaluated by accelerometer for 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Justina Kanold, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France